CLINICAL TRIAL: NCT03644732
Title: Atlas of Human Cognition by SEEG
Brief Title: Atlas of Human Cognition by SEEG (MAPCOG-SEEG)
Acronym: MAPCOG-SEEG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.357; 2017-A03248-45 (Other: ID RCB)
Record Dates: First submitted 2018-04-09; First posted 2018-08-23 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Refractory Epilepsy; Focal Epilepsy
Keywords: Cognition
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SEEG Group: Group with SEEG analysis (Pre-surgical SEEG assessment)
  Interventions: Procedure: SEEG Group

INTERVENTIONS:
Procedure: SEEG Group — Visual and quantitative SEEG signal analysis. As available, collection of behavioral and neuropsychological postsurgical data

SUMMARY:
The main objective of MAPCOG_SEEG is to create a database including brain recordings of cognition performed in clinical routine in patients during the pre-surgical SEEG assessment. This aims to be able to propose the first atlas of human cognition with a high temporal and spatial resolution.

DETAILED DESCRIPTION:
The pre-surgical assessment of a cortectomy in patient suffering from a refractory epilepsy includes several examinations aiming both, to specify the epileptogenic zone (EZ) which must be resected and to evaluate functional and cognitive risks of surgery.

Nevertheless, in some patients, non-invasive evaluation does not give formal answer. In these subjects, it is then necessary to carry out a second step, consisting of an invasive exploration by implantation of intracerebral electrodes during a Stereoelectroencephalography (SEEG).

Due to its temporal and spatial resolution, the SEEG allows, besides the precise determination of the EZ, to carry out a functional mapping of the cortical regions likely to be included in cortectomy. Conventionally, this mapping is carried out on the basis of the cortical electrical stimulations applied to the implanted electrodes. If this approach is very robust for exploring primary functions such as motor skills or language, it cannot be used to evaluate more complex cognitive tasks such as face recognition or attention. Essential cognitive tasks on a daily basis.

This has led to the development in recent years, in Grenoble, of a complementary approach to cerebral stimulation: Dynamic Spectral Imaging (ISD). Numerous experimental paradigms have demonstrated that the realization of a cognitive task associates with the generation within the cortical regions involved in its treatment of a particular cortical activity. This activity is characterized by oscillations of the cortical rhythm in high frequencies (> 40 Hz), called gamma activities. The ISD thus consists in mapping this gamma activity during various cognitive tasks, thus making it possible to study more widely the complexity of the cognitive functions.

MAPCOG_SEEG aims to collect the cerebral recording of the patients who have performed this cognitive exploration to be able to in fine propose an Atlas of human cognition which takes advantage of the very rich information in terms of spatial and temporal resolution of the SEEG. Furthermore, it will exactly allow more to understand the impact of the epilepsy and the surgery of the epilepsy on the cognition.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant focal epilepsy
* Justified SEEG exploration in the context of presurgical assessment of epilepsy
* Written non-opposition to study participation
* Intellectual capacities compatible with the compliance in the cognitive tasks

Exclusion Criteria:

* Major Patient undergoing a legal protection measure or patient deprived of liberty as a result of a judicial or administrative decision
* Impossibility of collecting information on exposure (recent arrival in France, foreign language, etc.)
* Pregnant women (Contraindication to SEEG exploration)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (Age between 18 and 65 years) patients receiving an SEEG exploration for presurgical evaluation of focal refractory epilepsy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
SEEG recordings using functional brain mapping procedure (composite measures) | 3 weeks
  Prospective collection of data from SEEG recordings using functional brain mapping procedure performed in clinical routine during the presurgical assessment of patients with drug-resistant epilepsy. These data are represented by the electroencephalographic activity during the realization of the different cognitive tasks proposed to the patients. Electroencephalographic activity will then be analyzed in terms of Dynamic Spectral Imaging and in terms of high frequency activity ([50-150Hz]).

SECONDARY OUTCOMES:
Behavioral data (composite measures) | 3 weeks
  Behavioral data (reaction time and accuracy of response) collected during the presurgical assessment (joint with the SEEG) and during the postsurgical follow-up (approximately 3 months after the surgery) as well as the collection of neuropsychological scores from the presurgical and postsurgical assessment.
  Behavioral performance and neuropsychological test scores before and after surgery (as available) will allow to evaluate the impact of surgery on cognitive functioning (improvement or deterioration of cognitive performance).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kahane, MD/PhD, Principal Investigator — University Hospital, Grenoble; Marcela Perrone-Bertolotti, PhD, Study Chair — Centre National de la Recherche Scientifique, France
Locations (4):
- France (4):
  - University Hospital, Grenoble, Grenoble
  - CHRU Nancy, Nancy
  - Hôpital Ste Anne, Paris
  - CHU Rennes, Rennes

REFERENCES:
- [Background] Lachaux JP, Axmacher N, Mormann F, Halgren E, Crone NE. High-frequency neural activity and human cognition: past, present and possible future of intracranial EEG research. Prog Neurobiol. 2012 Sep;98(3):279-301. doi: 10.1016/j.pneurobio.2012.06.008. Epub 2012 Jun 26. PMID 22750156
- [Result] Baciu M, Perrone-Bertolotti M. What do patients with epilepsy tell us about language dynamics? A review of fMRI studies. Rev Neurosci. 2015;26(3):323-41. doi: 10.1515/revneuro-2014-0074. PMID 25741734
- [Result] Combrisson E, Perrone-Bertolotti M, Soto JL, Alamian G, Kahane P, Lachaux JP, Guillot A, Jerbi K. From intentions to actions: Neural oscillations encode motor processes through phase, amplitude and phase-amplitude coupling. Neuroimage. 2017 Feb 15;147:473-487. doi: 10.1016/j.neuroimage.2016.11.042. Epub 2016 Nov 30. PMID 27915117
- [Result] Ossandon T, Vidal JR, Ciumas C, Jerbi K, Hamame CM, Dalal SS, Bertrand O, Minotti L, Kahane P, Lachaux JP. Efficient "pop-out" visual search elicits sustained broadband gamma activity in the dorsal attention network. J Neurosci. 2012 Mar 7;32(10):3414-21. doi: 10.1523/JNEUROSCI.6048-11.2012. PMID 22399764
- [Result] Perrone-Bertolotti M, Vidal JR, de Palma L, Hamame CM, Ossandon T, Kahane P, Minotti L, Bertrand O, Lachaux JP. Turning visual shapes into sounds: early stages of reading acquisition revealed in the ventral occipitotemporal cortex. Neuroimage. 2014 Apr 15;90:298-307. doi: 10.1016/j.neuroimage.2013.12.027. Epub 2013 Dec 24. PMID 24370818
- [Result] Perrone-Bertolotti M, Kujala J, Vidal JR, Hamame CM, Ossandon T, Bertrand O, Minotti L, Kahane P, Jerbi K, Lachaux JP. How silent is silent reading? Intracerebral evidence for top-down activation of temporal voice areas during reading. J Neurosci. 2012 Dec 5;32(49):17554-62. doi: 10.1523/JNEUROSCI.2982-12.2012. PMID 23223279